CLINICAL TRIAL: NCT03914339
Title: "EFFECT OF ORTHODONTIC TREATMENT ON PERIODONTAL HEALTH OF PERIODONTALLY COMPROMISED DENTITION- A Prospective Randomized Controlled Clinical Trial"
Brief Title: Effect of Orthodontic Treatment on Periodontally Compromised Dentition- Randomised Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: meenu ortho
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Orthodontics; Periodontal Index

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Eighteen periodontally compromised patients who will be given both orthodontic and periodontal treatment .
  Interventions: Procedure: Periodontal and orthodontic treatment
- control group (Active Comparator): Eighteen periodontally compromised patients will receive periodontal treatment alone .
  Interventions: Procedure: periodontal treatment

INTERVENTIONS:
Procedure: Periodontal and orthodontic treatment — Eighteen periodontally compromised patients who give be given both periodontal and orthodontic treatment
  Arms: Test group
Procedure: periodontal treatment — Eighteen periodontally compromised patients who give be given periodontal treatment alone.
  Arms: control group

SUMMARY:
The main aim of this prospective, randomized controlled clinical study is to:

• To evaluate and compare the effect of a combined orthodontic -periodontal treatment protocol versus periodontal treatment alone on osseous and non -osseous parameters in periodontally compromised patients.

DETAILED DESCRIPTION:
All the patients of both the groups will receive a detailed periodontal evaluation and then therapeutic management of patients will be done as per their periodontal requirement. This will include oral hygiene instruction, scaling and root planning and re-evaluation after 2 weeks and periodontal surgical treatment if indicated will be re-evaluated 4-6 weeks. After an observation period of 2 months confirming patient cooperation and their ability to maintain good oral hygiene as well as stability of the periodontal results orthodontic treatment will be started in the test group whereas the control group will be kept on monthly recall for the first 3 months and then every 3 months as per the oral hygiene status requirement of the patient.periodontal charting will be done at every 3 months till finish of treatment and supra gingival scaling will be provided as per requirement in both the groups.Changes in periodontal status in terms of clinical and radiographic parameters will be compared between the groups. cone beam Computed tomography will be taken at the baseline T0 and study end point T2 for assessment of changes in the bone level around maxillary and mandibular teeth

ELIGIBILITY:
Inclusion Criteria

.• Patient age criteria 20-40 years.

* Periodontally Compromised dentition with moderate to severe periodontitis ≥2 teeth with pocket depth (PD) ≥5 mm and loss of clinical attachment level (CAL) ≥ 4mm. and radiographic bone loss
* Good general health status.
* Malocclusion that needs orthodontic treatment

Exclusion Criteria:

* Systemic illness known to affect the periodontium or outcome of periodontal and orthodontic therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Pregnant or lactating women.
* Smokers(≥5 cigarettes∕ day).
* Noncompliance to oral hygiene measures after Phase I therapy.
* Presence of trauma from occlusion (TFO).
* Patients with aggressive periodontitis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
• Alveolar crest bone level | 12 months
  measured from Cemento- enamel junction to bone crest.
Clinical attachment level (CAL). | 12 months
  • pocket to cemento- enamel junction .

CONTACTS AND LOCATIONS:
Overall Officials: Rekha sharma, MDS, Study Chair — PGIDS,ROHTAK
Locations (2):
- India (2):
  - Pgids,Rohtak, Rohtak, Haryana
  - PGIDS, Rohtak, Haryana